CLINICAL TRIAL: NCT04446286
Title: Bicentric Study on the Use of ECMO-VV or VA for Severe ARDS Associated With Covid-19
Acronym: ECMO-SL-CoV-2
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7904
Record Dates: First submitted 2020-06-23; First posted 2020-06-24 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2020-06

CONDITIONS: Covid-19
Keywords: Respiratory Distress Syndrome; SARS-CoV-2; Extracorporeal membrane oxygenation; ECMO-VV; ECMO-VA; Veno-venous ECMO
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Describes the cohort of patients receiving ECMO-VV or ECMO-VA in the management of severe ARDS refractory to SARS-CoV-2 in the Strasbourg and Louvain centres

ELIGIBILITY:
Inclusion Criteria:

* Patient over the age of 18;
* Diagnostic COVID-19 by RT-PCR;
* Hospitalisation in resuscitation for the management of complications related to COVID-19
* Implanted ECMO-VV or VA during hospitalisation;
* Patient agreeing to participate in the study

Exclusion Criteria:

* Sujet who has expressed opposition to participating in the study.
* Sujet under guardianship or trusteeship
* Sujet under safeguard of justice

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with a COVID-19 diagnosis by RT-PCR
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2020-08-18 (Actual)

PRIMARY OUTCOMES:
Retrospective description of effect of the ECMO-VV or ECMO-VA in the management of severe ARDS refractory in patients of the Strasbourg and Louvain centres with covid-19 | files analysed retrospectily from March 1st, 2020 to August 1st, 2020 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie Thoracique Nouvel Hôpital Civil Hôpitaux Universitaires de Strasbourg, Strasbourg, France